CLINICAL TRIAL: NCT00902135
Title: Betaferon® Injection Management: Non-interventional Study on Personal Digital Assistant (PDA)Supported Effects on Adherence to a Long-term Injection Therapy (BETAPATH)
Brief Title: Injection Management With Betaferon: Influence on Adherence, Patients Satisfaction and Health Related Outcomes (BETAPATH)
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 14543; BF0801DE (Other: Company internal)
Record Dates: First submitted 2009-05-13; First posted 2009-05-14 (Estimated); Last update posted 2015-07-17 (Estimated); Status verified 2015-07

CONDITIONS: Relapsing-Remitting Multiple Sclerosis
Keywords: Multiple Sclerosis; Interferon beta-1b
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Interferon beta-1b

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Group 1
  Interventions: Drug: Interferon beta-1b (Betaseron, BAY86-5046)
- Group 2
  Interventions: Drug: Interferon beta-1b (Betaseron, BAY86-5046)
- Group 3
  Interventions: Drug: Interferon beta-1b (Betaseron, BAY86-5046)

INTERVENTIONS:
Drug: Interferon beta-1b (Betaseron, BAY86-5046) — Interferon beta-1b (Betaferon) and Personal Digital Assistant together with a reminder
  Groups: Group 1
Drug: Interferon beta-1b (Betaseron, BAY86-5046) — Interferon beta-1b (Betaferon) and Personal Digital Assistant without a reminder
  Groups: Group 2
Drug: Interferon beta-1b (Betaseron, BAY86-5046) — Interferon beta-1b (Betaferon)
  Groups: Group 3

SUMMARY:
Aim of the BETAPATH study is to evaluate whether the use of a personal digital assistant (PDA) can improve the adherence of Multiple Sclerosis patients to a therapy with Betaseron. The Personal digital assistant PDA functions as an electronic diary and as an injection reminder.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with the diagnosis of Multiple Sclerosis and decision by the investigator to prescribe Betaferon.The decision for treatment type and duration is taken before offering the patient the possibility to participate in the study.

Exclusion Criteria:

* Patients, who do not meet the Clinically Isolated Syndrome (CIS) or Relapsing/Remitting Multiple Sclerosis (RRMS) criteria, should not be included.
* Exclusion criteria must be read in conjunction with the German product information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult female and male Clinically Isolated Syndrome (CIS) and relapsing-remitting multiple sclerosis (RRMS) patients who are at least 18 years of age, have started a treatment with Betaferon based on clinical decision by the treating neurologist and have completed the dose titration, will be documented after the therapy decision has been made.
  The prescription of the medicine must be clearly independent from the decision to include the patient in the study.
Sampling Method: Non-Probability Sample
Enrollment: 702 (Actual)
Dates: Start 2009-05; Primary Completion 2013-12 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Drop out rate over 2 years | 24 months

SECONDARY OUTCOMES:
Disability status | After 3, 6, 12 and 24 months
Grade of depressiveness | After 3, 6, 12 and 24 months
Grade of fatigue | After 3, 6, 12 and 24 months
Quality of life | After 3, 6, 12 and 24 months
Cognitive status | After 12 and 24 months
Injection regularity | After 3, 6, 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Germany

REFERENCES:
- [Derived] Zettl UK, Bauer-Steinhusen U, Glaser T, Hechenbichler K, Hecker M; Study Group. Comparative evaluation of patients' and physicians' satisfaction with interferon beta-1b therapy. BMC Neurol. 2016 Sep 21;16(1):181. doi: 10.1186/s12883-016-0705-1. PMID 27653529
- [Derived] Zettl UK, Bauer-Steinhusen U, Glaser T, Czekalla J, Hechenbichler K, Limmroth V, Hecker M. Adherence to Long-Term Interferon Beta-1b Injection Therapy in Patients with Multiple Sclerosis Using an Electronic Diary. Adv Ther. 2016 May;33(5):834-47. doi: 10.1007/s12325-016-0325-6. Epub 2016 Apr 18. PMID 27090116
- [Derived] Zettl UK, Bauer-Steinhusen U, Glaser T, Hechenbichler K, Limmroth V; Study Group. Evaluation of an electronic diary for improvement of adherence to interferon beta-1b in patients with multiple sclerosis: design and baseline results of an observational cohort study. BMC Neurol. 2013 Sep 6;13:117. doi: 10.1186/1471-2377-13-117. PMID 24011220